CLINICAL TRIAL: NCT00447954
Title: A Phase II Study of Implants of Encapsulated Human NTC-201 Cells Releasing Ciliary Neurotrophic Factor (CNTF), in Participants With Visual Acuity Impairment Associated With Atrophic Macular Degeneration
Brief Title: A Study of an Encapsulated Cell Technology (ECT) Implant for Patients With Atrophic Macular Degeneration
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neurotech Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CNTF 2; NCT00277134 (obsolete NCT alias)
Record Dates: First submitted 2007-03-09; First posted 2007-03-15 (Estimated); Results first posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Nonexudative Age-Related Macular Degeneration, Unspecified Eye, Intermediate Dry Stage
Keywords: eye disease; retinal disorder; CNTF; AMD; Atrophic AMD
MeSH Terms: conditions — Eye Diseases; Retinal Diseases | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- 1 - High Dose (Experimental): Participant had surgically implanted high dose (NT-501-6A.02) CNTF-secreting NT-501 device which produced ~20 ng/device/day.
  Interventions: Combination Product: High Dose NT-501 implant
- 2 - Low Dose (Experimental): Participant had surgically implanted high dose (NT-501-6A.02) CNTF-secreting NT-501 device which produced ~5 ng/device/day.
  Interventions: Combination Product: Low Dose NT-501 implant
- 3 - Sham (Sham Comparator): Sham surgery procedure in which no device was implanted
  Interventions: Other: Sham

INTERVENTIONS:
Combination Product: High Dose NT-501 implant — High Dose NT-501
  Arms: 1 - High Dose
Combination Product: Low Dose NT-501 implant — Low Dose NT-501
  Arms: 2 - Low Dose
Other: Sham — Sham Procedure
  Arms: 3 - Sham

SUMMARY:
The purpose of this study is to look at the safety and effectiveness of CNTF implants on vision in participants with atrophic macular degeneration. This research is being done because there are no effective therapies for people with atrophic macular degeneration. Age-related macular degeneration (AMD) is a condition that affects the macula, the central part of the retina that we use for seeing details. There are two types of AMD, one is the wet type in which new blood vessels grow, also known as choroidal neovascularization (CNV), but the other is the dry type in which the healthy cells die, and that is the target of this study. This is called atrophic macular degeneration. The implant is a small capsule that contains human retinal pigment epithelium cells. These cells have been given the ability to make CNTF and release it through the capsule membrane into the surrounding fluid. In this study, two different CNTF dose levels will be used: a high dose and a low dose, as well as a sham surgery (or placebo) group.

DETAILED DESCRIPTION:
Histopathologic studies of multiple forms of retinal neurodegenerative diseases have demonstrated the possibility of using the neurotrophic factor CNTF as an effective approach to reducing photoreceptor cell loss. Consequently, it had been hypothesized that the use of the implanted NT-501 capsule, which secretes CNTF into the vitreous, might be beneficial in people with atrophic macular degeneration. The purpose of this pilot study was to accumulate preliminary data on the effect of the intraocular NT-501 implant on visual acuity in patients with atrophic macular degeneration.

The study had a double-masked, multi-center, randomized, parallel group design. Eligible patients were randomized on a 2:1:1 basis to the higher CNTF output NTC-201-6A.02 implant, the lower CNTF output NTC-201-10.02 implant or to sham surgery, respectively.

The surgeon designated by the Principal Investigator (PI), the PI, vision examiners, reading center graders, and patients were all masked as to the dose of the implant. The patients and the vision examiners were masked as to which treatment was received.

Approximately 48 patients with geographic atrophy compatible with category 3 or 4 AMD were planned to be enrolled. All patients were to be followed clinically for 18 months. Patients randomized to the CNTF implants were implanted at baseline, had the option of being explanted at or after 12 months, and all were followed clinically for 18 months. Follow-up for safety occurred throughout the study period.

ELIGIBILITY:
Study inclusion criteria:

1. To participate in this study, the participant had to understand and sign the protocol's informed consent (if the participant's vision was impaired to the point where it was not possible to read the informed consent document, the informed consent document was read in its entirety to the participant).
2. Women of childbearing potential (women with last menses <1 year prior to screening) had to agree to use an effective form of birth control from study onset until they completed the 18 month study visit.
3. Participant had to be medically able to undergo ophthalmic surgery for NT-501 implant.
4. Best-corrected visual acuity in the study eye between 20/50 and 20/200 (68-34 letter score) as measured using EVA.
5. Presence in the study and/or fellow eye of geographic atrophy (GA) compatible with category 3 or 4 age-related macular degeneration (AMD) as defined by AREDS (AREDS, 2001). Also, the GA in the study eye had to be associated with vision loss as assessed by a vision test. GA was defined as one or more well-defined, usually more or less circular patches of partial or complete depigmentation of the RPE, typically with exposure of underlying choroidal blood vessels. Even if much of the RPE appeared to be preserved and large choroidal vessels were not visible, a roundish patch of RPE partial depigmentation might still be classified as early GA. A patch had to be at least 175 microns in area.
6. Participants had steady fixation in the study eye in the foveal or parafoveal area with media clear enough for good quality photographs.

Study exclusion criteria:

1. Participant less than 50 years of age (to minimize geographic atrophy from causes other than AMD).
2. Participant medically unable to comply with study procedures or follow-up visits.
3. Participant had evidence of ocular disease other than AMD that might confound the outcome of the study (e.g., diabetic retinopathy, uveitis, etc.).
4. Participant had chronic requirement (e.g., > or = 4 weeks at a time) for ocular medications or had disease(s), that in the judgment of the examining physician, were vision threatening or might affect the primary outcome (artificial tears were permitted).
5. Participant had evidence of classic or occult choroidal neovascularization in either eye, which might include serous RPE detachment, stippling on a fluorescein angiogram, macular edema, evidence of hemorrhage and lipid, and disciform scar.
6. Participant had a requirement for acyclovir and/or related products during study duration. To be eligible for this study, the participant had to discontinue use of these products prior to enrollment and could not continue with the products until after they had completed the study.
7. Participant had evidence of central serous chorio-retinopathy (CSR) in either eye.
8. Participant had evidence of pathologic myopia in either eye.
9. Participant had evidence of pseudovitelliform macular degeneration (a dominantly inherited disease characterized by a round or oval yellow subretinal macular deposit) in either eye.
10. Participant was receiving systemic steroids or other immunosuppressive medications.
11. Participant with evidence of vitreo-retinal traction maculopathy in either eye.
12. Participant had a history of laser, photodynamic therapy (PDT), intravitreal injection of antivascular endothelial growth factor (VEGF) agent, or any previous treatment for AMD other than AREDS or equivalent supplement formulation.
13. Prior history of vitrectomy, penetrating keratoplasty, trabeculectomy or trabeculoplasty.
14. Participant had any of the following lens opacities: cortical opacity > standard 3, posterior subcapsular opacity > standard 3, or a nuclear opacity > standard 3 as measured on the AREDS clinical lens grading system.
15. Participant had undergone lens removal in the last 3 months.
16. Participant had participated in any other clinical trial of a drug or within the last 6 months.
17. Participant was on chemotherapy.
18. Participant was on ocular or systemic medications known to be toxic to the lens, retina, or optic nerve.
19. Participant was pregnant or lactating.
20. Participant had other retinal disease(s).
21. Participant had a history of malignancy, except study participants with a history of successfully treated cancer (≥5 years prior to inclusion in the trial).
22. Participant was considered immunodeficient or had a known history of HIV.
23. Participant with a history of ocular herpes zoster.
24. Participant's fellow eye visual acuity worse than 20/400.
25. Participant had undergone LASIK surgery or other refractive surgery for either eye in less than 6 months prior to screening.
26. Participants with severe hearing disabilities in both ears.
27. Participants with unmanaged diabetes, patients with CME, or retinopathy in either eye.
28. Participant had a history of retinal detachment in either eye.
29. Participant who had been diagnosed and treated for amblyopia as an infant.
30. Participant with a history of Pars Plana Vitrectomy.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2007-01-05 (Actual); Primary Completion 2009-05-11 (Actual); Study Completion 2009-05-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Weng Tao, M.D., PhD, Study Director — Neurotech Pharmaceuticals
Locations (8):
- United States (8):
  - Retina-Vitreous Associates Medical Group, Beverly Hills, California
  - Retina Group of Florida, Hollywood, Florida
  - Bascom Palmer Eye Institute, Miami, Florida
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - Beaumont Eye Institute, Royal Oak, Michigan
  - Retina Foundation of Southwest, Dallas, Texas
  - Vitreoretinal Consultants, Houston, Texas
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kauper K, McGovern C, Sherman S, Heatherton P, Rapoza R, Stabila P, Dean B, Lee A, Borges S, Bouchard B, Tao W. Two-year intraocular delivery of ciliary neurotrophic factor by encapsulated cell technology implants in patients with chronic retinal degenerative diseases. Invest Ophthalmol Vis Sci. 2012 Nov 1;53(12):7484-91. doi: 10.1167/iovs.12-9970. PMID 23049090

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study had a double-masked, multi-center, randomized, parallel group design. Patients were randomized on a 2:1:1 basis to the higher CNTF output NTC-201-6A.02 implant, the lower CNTF output NTC-201-10.02 implant or to sham surgery. A total of 53 patients were randomized to the treatment groups: 27 patients to the higher CNTF output NTC-201-6A.02 implant, 13 patients to the lower CNTF output NTC-201-10.02 implant and 13 patients to sham surgery.
Pre-assignment Details: Two patients withdrew following randomization but prior to the implantation/sham surgery procedure (one in the low-output implant arm and one in the sham surgery arm).
  Four patients withdrew early, all in the high dose treatment group. In two cases, withdrawal was due to AEs; one patient was lost to follow up and one withdrew consent.
Units Other Than Participants: Eyes
Groups:
- Low Dose: NT-501 implant: Low Dose encapsulated cell therapy that delivers ciliary neurotrophic factor to the retina
- High Dose: NT-501 implant: High Dose encapsulated cell therapy that delivers ciliary neurotrophic factor to the retina
- Sham: No implant (Sham procedure)
  Non-penetrating sham procedure to mimic implant procedure
Period: Overall Study
Arm/Group | Low Dose | High Dose | Sham
Started | 13; 13 Eyes | 27; 27 Eyes | 13; 13 Eyes
Completed | 12; 12 Eyes | 23; 23 Eyes | 12; 12 Eyes
Not Completed | 1; 1 Eyes | 4; 4 Eyes | 1; 1 Eyes
Not completed — Adverse Event | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Exclusionary event prior to implant procedure | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants who were randomized to a study arm but prior to surgical procedure.
Units Other Than Participants: eyes
Groups:
- Low Dose: NT-501 implant: Low Dose
- High Dose: NT-501 implant: High Dose
- Sham: No implant (Sham Procedure)
- Total: Total of all reporting groups
Arm/Group | Low Dose | High Dose | Sham | Total
Number analyzed (Participants) | 13 | 27 | 13 | 53
Number analyzed (eyes) | 13 | 27 | 13 | 53
Age, Continuous [Mean (Standard Deviation); unit: Years] | 78.3 (5.6) | 74.9 (7.5) | 74.5 (6.0) | 75.6 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 17 | 5 | 28
  Male | 7 | 10 | 8 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 13 | 27 | 13 | 53
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 13 | 27 | 13 | 53
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Ocular History [Mean (Standard Deviation); unit: Years] — Baseline measures were assessed for all randomized participants (13 - Low Dose, 27 - High Dose, 13 - Sham).
  Years
    Years since first diagnosed with AMD | 6.75 (6.81) | 8.39 (6.82) | 9.84 (9.06) | 8.34 (7.36)
    Years since ocular disease | 2.89 (3.54) | 3.44 (4.34) | 5.93 (9.63) | 3.92 (5.92)
    Years since ocular surgery | 5.99 (6.13) | 4.73 (4.31) | 2.49 (1.66) | 4.65 (4.64)
    Years since ocular treatment | 1.60 (0.0) | 5.18 (3.68) | 2.63 (0.0) | 3.65 (2.79)
Type of Ocular History [Number; unit: Participants]
  Ocular Disease | 13 | 27 | 13 | 53
  Ocular Surgery | 9 | 13 | 6 | 28
  Ocular Treatment | 1 | 2 | 1 | 4
Baseline BCVA [Mean (Standard Deviation); unit: Letter score (# of letters read correct)] — Monocular Best Corrected Visual Acuity (BCVA), assessed by eye for each participant. Population: N=number of eyes assessed in all treated participants (mITT population)
  Letter score (# of letters read correct)
    number analyzed (Participants) | 12 | 27 | 12 | 51
    Treated Eye | 49.9 (10.2) | 53.5 (9.0) | 56.3 (6.6) | 53.2 (8.6)
    Untreated Eye | 55.7 (23.2) | 55.0 (21.6) | 68.1 (9.1) | 59.6 (18.0)

OUTCOME MEASURES:

1. Primary Outcome: BCVA Response Defined as an Increased in 10 Letters at 1 Year Post-implant
Description: Response is defined as a improvement from baseline at Month 12 in monocular best visual acuity (BCVA) in the study eye of at least 10 letters as assessed by standard Early Treatment Diabetic Retinopathy Study (ETDRS) chart.
Time Frame: 1 year post-implant
Population: N=number of eyes assessed in all treated participants (mITT population)
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Low Dose | High Dose | Sham
Number analyzed (Participants) | 12 | 27 | 12
Number analyzed (eyes) | 12 | 27 | 12
eyes
  Response | 3 | 3 | 1
  No Response | 9 | 24 | 11

2. Secondary Outcome: The Change in BCVA Over the 18-month Follow-up Period
Description: Change from baseline at post-baseline visits in monocular best visual acuity (BCVA) as assessed by standard Early Treatment Diabetic Retinopathy Study (ETDRS) chart.
Time Frame: From initial implant 18 months post-implant
Population: N=number of eyes assessed in all treated participants (mITT population)
Measure: Mean (Standard Deviation); unit: Letter score (number of letters)
Units Other Than Participants: eyes
Arm/Group | Low Dose | High Dose | Sham
Number analyzed (Participants) | 12 | 27 | 12
Number analyzed (eyes) | 12 | 27 | 12
Letter score (number of letters)
  1 month post-implant - Treated | -0.1 (6.6) | 1.5 (5.5) | 1.4 (6.2)
  1 month post-implant - Untreated | 1.0 (6.1) | 2.9 (6.5) | 0.5 (3.1)
  3 months post-implant - Treated | -4.4 (7.9) | 3.0 (4.7) | 2.1 (8.8)
  3 months post-implant - Untreated | -0.5 (4.4) | 2.3 (6.1) | -0.5 (6.7)
  4 months post-implant - Treated | -0.8 (11.2) | 3.0 (5.9) | 2.9 (7.7)
  4 months post-implant - Untreated | -1.0 (5.4) | 2.9 (7.2) | 0.3 (7.3)
  6 months post-implant - Treated: number analyzed (Participants) | 12 | 26 | 12
  6 months post-implant - Treated | -0.1 (11.8) | 2.7 (5.3) | -0.4 (7.7)
  6 months post-implant - Untreated: number analyzed (Participants) | 12 | 26 | 12
  6 months post-implant - Untreated | -1.6 (9.3) | 1.5 (7.7) | -1.9 (6.1)
  12 months post-implant - Treated | -0.3 (15.9) | -0.2 (8.4) | -1.3 (11.1)
  12 months post-implant - Untreated | -4.6 (17.9) | -1.8 (14.4) | -6.0 (9.6)
  18 months post-implant - Treated: number analyzed (Participants) | 10 | 21 | 12
  18 months post-implant - Treated | -1.8 (18.4) | -5.3 (15.0) | -4.1 (13.7)
  18 months post-implant - Untreated: number analyzed (Participants) | 10 | 21 | 12
  18 months post-implant - Untreated | -7.0 (14.6) | -3.7 (13.5) | -8.5 (11.1)

ADVERSE EVENTS:
Time Frame: All patients were to be followed clinically for 18 months. Patients could have the implant removed (explanted) from the eye after 12 months or earlier in case of adverse events (AEs) or at the patient's request. Patients were followed up to 18-months post implant.
Description: No serious adverse events or study withdrawals related to the implantation procedure or the active study treatment. Although all patients experienced at least one AE during the study period, the majority were mild or moderate in severity. No severe or life-threatening AEs were considered to be related to the study treatments or study procedures.
  One SAE (cardiac arrest experienced by a patient in the high dose group) resulted in death. There were no other deaths during the study.
Arm/Group | Low Dose | High Dose | Sham
All-Cause Mortality (participants affected / at risk) | 0/12 | 1/27 | 0/12
Serious Adverse Events (participants affected / at risk) | 1/12 | 10/27 | 1/12
Other Adverse Events (participants affected / at risk) | 4/12 | 8/27 | 2/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose (N=12) | High Dose (N=27) | Sham (N=12)
Acute Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Choriodal Neovascularisation (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Retinal Haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis Radiation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Hip Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Metastatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Carotid Artery Occlusion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Mental Status Change (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Postmenopausal Haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral Arterial Occlusive Disease (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral Ischaemia (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose (N=12) | High Dose (N=27) | Sham (N=12)
Anterior Chamber Cell (Eye disorders) | 1 (1) | 2 (2) | 0 (0)
Anterior Chamber Flare (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Cataract Cortical (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Cataract Subcapsular (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Conjuctival Haemorrhage (Eye disorders) | 0 (0) | 3 (3) | 0 (0)
Conjunctival Hyperaemia (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
Eye Discharge (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Eye Irritation (Eye disorders) | 0 (0) | 2 (2) | 1 (1)
Eye Pain (Eye disorders) | 1 (1) | 2 (2) | 1 (1)
Eye Pruritis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Eyelid Ptosis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Lacrimation Increased (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Miosis (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Ocular Hyperaemia (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Photopsia (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Retinal Haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Visual Disturbance (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Vitreous Disorder (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Vitreous Haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Eye Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Suture Related Complication (Injury, poisoning and procedural complications) | 0 (0) | 4 (4) | 0 (0)
Intraocular Pressure Increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes